CLINICAL TRIAL: NCT03681964
Title: Diagnostic Suspicion of Primitive Syndrome Sjögren's : Brest Cohort
Acronym: DIApSS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: DIApSS
Record Dates: First submitted 2018-09-21; First posted 2018-09-24 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-07

CONDITIONS: Primary Sjögren's Syndrome (pSS)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to evaluate the diagnosis performance of several item used for the classification, the diagnosis and the prognostic of pSS (primary Sjogren syndrome)

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected pSS underwent a standardised evaluation

Exclusion Criteria:

* Opposition of patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected pSS underwent a standardised evaluation
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09-28 (Actual); Primary Completion 2020-09-28 (Estimated); Study Completion 2030-09-28 (Estimated)

PRIMARY OUTCOMES:
classification criteria | Inclusion (Day 0)
  classification criteria at inclusion of patients with suspected primary Sjögren's syndrome (pSS) underwent with standardised evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Devauchelle, Study Director — CHRU de Brest
Locations (1):
- CHRU de Brest, Brest, France